CLINICAL TRIAL: NCT00869115
Title: A Randomized, Double-blind, Placebo-controlled Escalating Dose Phase I Interaction Study to Evaluate the Pharmacokinetics, Tolerability and Pharmacodynamics of Three Dose Levels of Debio 0614 (Istaroxime) as a 24-hour Constant Rate IV Infusion in Combination With Chronic Oral Digoxin Treatment in Patients With Controlled Cardiac Failure and Decreased Left Ventricular Systolic Function
Brief Title: Phase I Interaction Study of Istaroxime and Digoxin in Subjects With Stable Heart Failure
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was not started due to a re-evaluation of the istaroxime development program
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Hein Van Ingen, Medical Director, Debiopharm S.A.
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Debio 0614-106; PAREXEL Study Number : 98378
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Heart Failure
Keywords: Digoxin; Inotropes; Lusitropic agents; Istaroxime; Debio 0614
MeSH Terms: conditions — Heart Failure | interventions — Istaroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): TREATMENT 0.5 μg/kg/min
  Interventions: Drug: Istaroxime
- 2 (Experimental): TREATMENT 1.0 μg/kg/min
  Interventions: Drug: Istaroxime
- 3 (Experimental): TREATMENT 1.5 μg/kg/min
  Interventions: Drug: Istaroxime
- 4 (Placebo Comparator): PLACEBO
  Interventions: Drug: Istaroxime

INTERVENTIONS:
Drug: Istaroxime — Istaroxime 0.5 μg/kg/min (30 μg/kg/h) continuous i.v. infusion for 24 hours
  Arms: 1
Drug: Istaroxime — Istaroxime 1.0 μg/kg/min (60 μg/kg/h) continuous i.v. infusion for 24 hours
  Arms: 2
Drug: Istaroxime — Istaroxime 1.5 μg/kg/min (90 μg/kg/h) continuous i.v. infusion for 24 hours
  Arms: 3
Drug: Istaroxime — Placebo continuous i.v. infusion for 24 hours
  Arms: 4

SUMMARY:
This study explores a potential drug-drug interaction between istaroxime and digoxin in patients with stable CHF on chronic oral digoxin treatment.

DETAILED DESCRIPTION:
This is a single center, randomized, double blind, placebo controlled, escalating dose phase I interaction study. The three dose levels of istaroxime or placebo will be randomized sequentially to three cohorts (I to III) of 16 patients each (12 patients on istaroxime and 4 patients on placebo). Digoxin will be administered non blinded in all patients, once daily in the morning after a standardized breakfast, continuing with previously personalized dosage schedule during the screening period, treatment period, post treatment period and follow up period. Prior to accrual of cohorts II and III, a Data Monitoring Committee (DMC) will advise on the continuation to the next istaroxime dose, based on a predetermined safety review.

This 37 day study includes a screening period (Days -21 to -1), a treatment period (Day 1), a post treatment period (Days 2-4), and a follow up period (which includes one patient visit on Day 14). Patients will be confined in the phase I research center from Day -2 to Day 4.

ELIGIBILITY:
Inclusion Criteria:

Main screening inclusion criteria :

* Signed informed consent;
* Male or female patients ≥18 years;
* Female patients of childbearing potential must not be pregnant;
* Chronic stable cardiac function impairment (no change in heart failure medication over the last 3 months and without any dosage adjustment in the last 4 weeks);
* Systolic blood pressure (SBP) of ≥ 90 mmHg and ≤ 140 mmHg;
* LVEF ≤ 35% by any method (to be performed at screening if not measured within the last 12 months);
* Chronic treatment (i.e. once daily dosing without interruption) with oral digoxin started at least 3 months prior to study entry and without any concomitant administration of other positive inotropic drugs;

Exclusion Criteria:

Main screening exclusion criteria :

* Need for current or intermittent intravenous positive inotrope administration within the preceding 6 months, or hemodynamic support devices;
* Acute coronary syndrome within the past 3 months;
* Coronary artery bypass graft or percutaneous coronary intervention within the past 3 months;
* Stroke within the past 6 months;
* Atrial fibrillation or uncontrolled heart rate (HR) (> 100 beats per minute [bpm]);
* Significant arrhythmia or second or third degree atrio-ventricular block;
* Valvular disease as the primary cause of HF;
* Significant ECG abnormalities as assessed by appropriately qualified physician or investigator including QTcF >450;
* Positive testing for Human Immunodeficiency Virus (HIV), Hepatitis B and/or Hepatitis C;

Main randomization exclusion criteria:

* HR > 100 bpm or < 50 bpm;
* Serum potassium > 5.3 mmol/L or < 3.8 mmol/L and magnesium > 1.1 mmol/L or < 0.6 mmol/L,
* TN I > ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Pharmacokinetic endpoints : Istaroxime PK parameters: - Istaroxime and Istaroxime metabolites (PST2915/2922/3093) plasma concentrations - Istaroxime and Istaroxime metabolites (PST2915/2922/3093) urine concentrations
Pharmacokinetic endpoints : Digoxin PK parameters: - Digoxin plasma concentrations
Safety endpoints: - Incidence of adverse events; - Change in vital signs; - Change in 12-lead ECG parameters; - Incidence of clinically or hemodynamically significant episodes of supraventricular or ventricular arrhythmias detected by continuous EC
Pharmacodynamic endpoints: - Change in echocardiographic parameters; - Change in SBP; - Change in non invasive cardiac output (Impedance cardiography) parameters.

REFERENCES:
- [Background] Gheorghiade M, Blair JE, Filippatos GS, Macarie C, Ruzyllo W, Korewicki J, Bubenek-Turconi SI, Ceracchi M, Bianchetti M, Carminati P, Kremastinos D, Valentini G, Sabbah HN; HORIZON-HF Investigators. Hemodynamic, echocardiographic, and neurohormonal effects of istaroxime, a novel intravenous inotropic and lusitropic agent: a randomized controlled trial in patients hospitalized with heart failure. J Am Coll Cardiol. 2008 Jun 10;51(23):2276-85. doi: 10.1016/j.jacc.2008.03.015. Epub 2008 Apr 9. PMID 18534276
- See also: Related Info — http://www.debiopharm.com